CLINICAL TRIAL: NCT03702361
Title: Rapid Intravenous Infusion of Velaglucerase Alfa (VPRIV) in Treatment-naive Patients With Type 1 Gaucher Disease: An Investigator-initiated Study
Brief Title: Rapid Intravenous Infusion of Velaglucerase Alfa (VPRIV) in Treatment-naive Patients With Type 1 Gaucher Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Ari Zimran, Professor, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-17-SZMC
Record Dates: First submitted 2018-08-06; First posted 2018-10-11 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Primary Disease
MeSH Terms: interventions — Glucosylceramidase

STUDY DESIGN:
Intervention Model Description: A single-center, open-label trial to assess the safety and efficacy of rapid administration of velaglucerase alfa (VPRIV) to treatment-naive patients with type I Gaucher disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapid infusion of Vpriv (Experimental): Rapid intravenous infusion of velaglucerase alfa (VPRIV) in treatment-naive patients with type 1 Gaucher disease
  Interventions: Drug: VPRIV

INTERVENTIONS:
Drug: VPRIV — VPRIV (Velaglucerase alfa) Long-term enzyme replacement therapy (ERT) for patients with type 1 Gaucher disease.
  Other Names: Velaglucerase Alfa

SUMMARY:
During the past two years, the investigator has performed succsefully an IIR wherein patients with GD, previously treated with velaglucerase alfa ERT were gradually switched to a 10 minutes (rapid) administration of the same ERT. The success was expressed as safety (no clinically meaningful AEs, no antibodies detected, home therapy), efficacy ("lack of deterioration") and patients' satisfaction. The latter was based not just on specific questionnaires and analog scales, but particularly by the patients' sharing the experience with other patients and consequently repeated requests by many to switch to a rapid administration of their ERT.

Therefore, the investigator is hereby proposing to investigate the safety and efficacy of a 10 minutes administration of velaglucerase alfa in a cohort of treatment-naive patients.

The current VPRIV label is restricted to a dosage of 60 units/kg body weight every other week (60 units/kg EOW) - this dose will be used throughout the study period. The enzyme will be provided by Shire, which will also provide a research grant for the conduction of the trial.

DETAILED DESCRIPTION:
Protocol:

Study Design: This will be a single-center, open-label trial to assess the safety and efficacy of rapid administration of velaglucerase alfa (VPRIV) to treatment-naive patients with type I Gaucher disease. The first six infusions will be administered in the hospital: the first three infusions within 60, 30 and 20 minutes each, with the beginning of a 10 minutes administration from infusion #4. Following the three uneventful administration of the 10 minutes in the hospital, the bi-weekly ERT will continue as home therapy, as outlined in the protocol. The duration of the study will be 12 months, with an extension pending positive results.

Number of Patients: 15. The first ten patients will be adults, and then children will be allowed to enroll in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years or older for the first ten adult patients; 6 years or older for the last five patients.

  * Confirmed enzymatic diagnosis of Gaucher disease with a defined genotype and elevated biomarker LysoGb1, performed at CentoGene using DBS methodology.
  * Indications for ERT will be guided by fulfilling the MOH criteria.
  * Female patients of child-bearing potential who agree to use a medically acceptable method of contraception.
  * Patients who have not received ERT or SRT in the past or Patients who have not received ERT or SRT in the past 12 months and have a negative anti-glucocerebrosidase antibody

Exclusion Criteria:

* Currently taking another experimental drug for any condition

  * Presence of neurologic signs and symptoms characteristic of Type 2 or Type 3 Gaucher disease
  * Pregnant or nursing
  * Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the patient's compliance with the study.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in spleen volume measured by MRI | 12 months.
  Percent change from baseline

SECONDARY OUTCOMES:
Change from baseline in Hemoglobin | 12 months
  Percent change from baseline
Change from baseline in platelet count | 12 months
  Percent change from baseline
Change from baseline in Lyso-GB1 | 12 months
  Percent change from baseline
Change from baseline in liver volume | 12 months
  Percent change from baseline
Change from baseline 10% reduction in spleen volume | 6 months
  Percent change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ari Zimran, M.D., Principal Investigator — Ari Zimran - Shaare Zedek
Locations (1):
- Michal Becker- Cohen, Jerusalem, Please Select..., Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zimran A, Revel-Vilk S, Becker-Cohen M, Chicco G, Arbel N, Rolfs A, Szer J. Rapid intravenous infusion of velaglucerase-alfa in adults with type 1 Gaucher disease. Am J Hematol. 2018 Sep;93(9):E246-E248. doi: 10.1002/ajh.25205. Epub 2018 Aug 9. No abstract available. PMID 29989200